CLINICAL TRIAL: NCT03640624
Title: Multidisciplinary Treatment of Chronic Vulvar Pain - a Randomized Controlled Study
Brief Title: Multidisciplinary Treatment of Chronic Vulvar Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016/2150
Record Dates: First submitted 2018-07-05; First posted 2018-08-21 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Vulvodynia; Chronic Pain
Keywords: Physical Therapy Modalities
MeSH Terms: conditions — Vulvodynia; Chronic Pain | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Multidisciplinary treatment
  Interventions: Combination Product: Multidisciplinary treatment
- Control (Active Comparator): Treatment as usual
  Interventions: Combination Product: Treatment as usual

INTERVENTIONS:
Combination Product: Multidisciplinary treatment — 1. Assessment by gynaecologist and dermatologist, resulting in tailored vulvar care, including daily topical lidocaine 5% ointment. Other topical or oral medication, such as oestradiol cream or oral antidepressants will be prescribed on individual basis.
  2. Tailored physiotherapy targeting muscular dysfunction, utilizing: Patient education, pelvic floor muscle exercises (contraction and relaxation), EMG-biofeedback. Low frequent electrical stimulation, massage, stretching and myofascial release and trigger point treatment of the pelvic floor. Desensitization exercises (manually or vaginal dilator). Relaxation and body awareness. Minimum one visit per month.
  3. Guided imagery sessions, minimum twice a week using a sound track that is developed for vulvodynia patients.
  Arms: Intervention
Combination Product: Treatment as usual — Treatment as usual in accordance with local guidelines by specialist in gynaecology, including a minimum of two visits (when diagnosis is made and after 3 - 6 months)
  Arms: Control

SUMMARY:
Vulvodynia (i.e. chronic vulvar pain without identifiable cause) is a heterogeneous clinical entity with a complex multifactorial causation. It is long lasting and difficult to treat, and the general consensus of current guidelines states that patients with vulvodynia benefit from a compound multidisciplinary intervention targeting mucosal hypersensitivity, pelvic muscle floor dysfunction and general pain management. However, there is little empiric evidence to support this recommendation. This will be a randomized controlled trial comparing multidisciplinary treatment with standard care for women with vulvodynia.

DETAILED DESCRIPTION:
Patients with chronic vulvar pain constitute a heterogeneous group with regards to causes and moderators of pain. Multidisciplinary teams simultaneously assess contributing factors such as infections and dermatoses and treat known mediators of pain, namely mucosal hypersensitivity, pelvic muscle floor dysfunction and general pain management. Treatment as usual, on the other hand, is primarily based on a sequential model applying one type of treatment at a time.

The investigator's aim is to compare multidisciplinary treatment including multimodal physiotherapy (intervention group) with standard treatment (control group) in reducing pain, sexual dysfunction and related symptoms in women with vulvodynia.

The study sample will be allocated randomly 1:1 to multidisciplinary treatment by a vulva team or to standard treatment by a specialist in gynaecology. The intervention will include a joint consultation by a gynaecologist and a dermatologist, tailored multimodal physiotherapy by a physiotherapist and guided imagery (mindfulness and relaxation) by use of a sound track during home sessions. The controls will receive standard care by a gynaecologist, who is free to offer any kind of non-standardized treatment.

Treatment effect will be measured at 3 months and at 6-12 months after inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years and older
* Chronic vulvar pain for ≥3 months of duration

Exclusion Criteria:

* Insufficient Norwegian skills
* Intellectual disability or severe mental disorder
* Severe comorbidity making tailored care necessary (such as active cancer treatment)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2024-11-10 (Actual); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Pain intensity with Brief pain inventory (BPI) | Baseline, 3 months and 6 months (change)
  Intensity of pain measured with BPI using the mean of the 4 subscales (current, averaged, maximum and minimum pain during the last week) on a 0-10 numerical rating scale (0 minimum and 10 maximum pain)

SECONDARY OUTCOMES:
Pain intensity with Brief pain inventory (BPI) | Baseline, 3 months, 6 months and 12 months (change)
  Intensity of pain measured with BPI using the mean of the 4 subscales (current, averaged, maximum and minimum pain during the last week) on a 0-10 numerical rating scale (0 minimum and 10 maximum pain)
Pain intensity with tampon test | Baseline and 6 months (change)
  Intensity of pain with tampon insertion and removal (tampon test) measured on a 0-10 numerical rating scale (0 minimum and 10 maximum pain)
Pain intensity with tampon test | Baseline, 6 months and 12 months (change)
  Intensity of pain with tampon insertion and removal (tampon test) measured on a 0-10 numerical rating scale (0 minimum and 10 maximum pain)
Vulvar pressure pain threshold with vulvalgesiometer | Baseline and 6 months (change)
  Vulvar pressure pain threshold in Newton measured with a cotton tipped vulvalgesiometer
Vulvar pressure pain threshold with vulvalgesiometer | Baseline, 6 months and 12 months (change)
  Vulvar pressure pain threshold in Newton measured with a cotton tipped vulvalgesiometer
Pain intensity with Short-Form McGill Pain Questionnaire-2 (SF-MPQ-2) | Baseline and 6 months (change)
  Pain intensity measured by a 22-Item NRS-based (0-10) questionnaire (SF-MPQ-2). Both total and subscale (continuous, intermittent, neuropathic, and affective pain) mean scores.
Pain intensity with Short-Form McGill Pain Questionnaire-2 (SF-MPQ-2) | Baseline, 6 months and 12 months (change)
  Pain intensity measured by a 22-Item NRS-based (0-10) questionnaire (SF-MPQ-2). Both total and subscale (continuous, intermittent, neuropathic, and affective pain) mean scores.
Sexual distress with Female Sexual Distress Scale - revised (FSDS) | Baseline and 6 months (change)
  Sexual distress measured with a 13-item Likert scale-based (0-4) questionnaire (FSDS). Mean score.
Sexual distress with Female Sexual Distress Scale - revised (FSDS) | Baseline, 6 months and 12 months (change)
  Sexual distress measured with a 13-item Likert scale-based (0-4) questionnaire (FSDS). Mean score.
Affective symptoms with Hospital Anxiety and Depression Scale (HADS) | Baseline and 6 months (change)
  Affective symptoms measured with a 14-item Likert scale-based (0-3) questionnaire (HADS). Both total and subscale (depression and anxiety) scores.
Affective symptoms with Hospital Anxiety and Depression Scale (HADS) | Baseline, 6 months and 12 months (change)
  Affective symptoms measured with a 14-item Likert scale-based (0-3) questionnaire (HADS). Both total and subscale (depression and anxiety) scores.
Illness perception with Brief Illness Perception Questionnaire (BIPQ) | Baseline and 6 months (change)
  Illness perception measured with a 8-Item NRS-based (0-10) questionnaire. Mean score of total scale.
Illness perception with Brief Illness Perception Questionnaire (BIPQ) | Baseline, 6 months and 12 months (change)
  Illness perception measured with a 8-Item NRS-based (0-10) questionnaire. Mean score of total scale.
Pain catastrophizing with Pain Catastrophizing Scale (PCS) | Baseline and 6 months (change)
  Pain catastrophizing measured with a 13-Item Likert scale-based (0-4) questionnaire (PCS). Total score.
Pain catastrophizing with Pain Catastrophizing Scale (PCS) | Baseline, 6 months and 12 months (change)
  Pain catastrophizing measured with a 13-Item Likert scale-based (0-4) questionnaire (PCS). Total score.
Levator hiatal area | Baseline and 6 months (change)
  Ultrasound-measured difference in levator hiatal area (cm^2) between rest and contraction and between rest and valsalva maneuver
Levator hiatal area | Baseline, 6 months and 12 months (change)
  Ultrasound-measured difference in levator hiatal area (cm^2) between rest and contraction and between rest and valsalva maneuver

CONTACTS AND LOCATIONS:
Overall Officials: Berit Schei, prof, Study Chair — Norwegian University of Science and Technology
Locations (1):
- Cecilie Hagemann, Trondheim, Norway